CLINICAL TRIAL: NCT02769936
Title: The Effects of D-cycloserine on Neuroplasticity and Working Memory in Healthy Adults and Patients With Schizophrenia
Brief Title: Glutamate, Learning, and Working Memory
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Robert F. Asarnow, Ph.D, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-000409
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia
Keywords: Receptors; N-Methyl-D-Aspartate
MeSH Terms: conditions — Schizophrenia | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Adult - Placebo (Placebo Comparator): Single dose placebo pill in healthy adults
  Interventions: Other: Placebo
- Healthy Adult - D-cycloserine (Experimental): Single 100 mg dose D-cycloserine pill in healthy adults
  Interventions: Drug: D-cycloserine
- Schizophrenia - Placebo (Placebo Comparator): Single dose placebo pill in schizophrenia patients
  Interventions: Other: Placebo
- Schizophrenia - D-cycloserine (Experimental): Single 100 mg dose D-cycloserine pill in schizophrenia patients
  Interventions: Drug: D-cycloserine

INTERVENTIONS:
Drug: D-cycloserine — 100 mg D-cycloserine administered orally as encapsulated pill
  Arms: Healthy Adult - D-cycloserine; Schizophrenia - D-cycloserine
Other: Placebo — Placebo administered orally as encapsulated pill
  Arms: Healthy Adult - Placebo; Schizophrenia - Placebo

SUMMARY:
Impairments in plasticity and working memory in schizophrenia have been hypothesized to reflect dysfunction at the N-methyl-D-aspartate glutamate receptor (NMDAR). However, the specific mechanisms through which the NMDAR is involved in working memory versus plasticity differ. Towards gaining a deeper understanding of how NMDAR signaling relates to individual cognitive functions in healthy adults and patients with schizophrenia, the investigators used a single dose of d-cycloserine (DCS) as an experimental probe to examine the effects of enhancing NMDAR signaling on plasticity versus working memory in healthy adults and individuals with schizophrenia.

DETAILED DESCRIPTION:
Background: Cognitive impairments in schizophrenia, such as deficits in plasticity and working memory, have been hypothesized to reflect dysfunction at the N-methyl-D-aspartate glutamate receptor (NMDAR). However, given that divergent properties of the NMDAR underlie its roles in plasticity versus working memory and that various aspects of NMDAR function are abnormal in schizophrenia, examining the effects of DCS in both healthy and patient populations is crucial.

Methods: The investigators used a single dose of the partial NMDAR agonist, d-cycloserine (DCS) to probe the effects of enhancing NMDAR signaling on working memory and plasticity. Working memory was assessed using a spatial n-back task. Plasticity was assessed using two learning tasks, the weather prediction task and information integration task, and an EEG paradigm that assesses changes in visual evoked potential amplitude following high frequency visual stimulation. Sixty-five healthy adults and forty-five schizophrenia patients were randomized to receive 100 mg acute DCS (healthy adult n = 32; schizophrenia n = 24) or placebo (healthy adult n = 33; schizophrenia n = 21).

ELIGIBILITY:
Inclusion criteria for healthy subjects:

1. between the ages of 18 and 30 years
2. comfortable reading in English
3. normal visual acuity or corrected vision
4. normal or corrected hearing.

Exclusion criteria for healthy subjects:

1. history or seizures or neurologic diseases
2. currently prescribed medication for any psychiatric conditions
3. any medical condition affecting fine motor movement of the hands
4. pregnancy or suspected pregnancy
5. use of recreational drugs or drugs taken not as prescribed in the past month
6. having a full scale intelligence quotient (IQ) < 70, as assessed by the Wechsler Abbreviated Scale of Intelligence (WASI)
7. having consumed alcohol in the 24 hours prior to the first lab visit
8. known allergy to any antibiotics.

Inclusion criteria for patients with schizophrenia:

1. between the ages of 18 and 50 years
2. comfortable reading in English
3. normal visual acuity or corrected vision
4. normal or corrected hearing
5. meets criteria for Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) diagnosis of schizophrenia.

Exclusion criteria for patients with schizophrenia:

1. history or seizures or neurologic diseases
2. currently prescribed Clozapine or medications contraindicated for DCS
3. any medical condition affecting fine motor movement of the hands
4. pregnancy or suspected pregnancy
5. history of traumatic brain injury requiring hospitalization for 2 or more days
6. IQ < 70, as assessed by the WASI
7. having consumed drugs other than as prescribed in the 48 hour prior to the testing visit or having consumed alcohol in the 24 hours prior to the testing visit
8. known allergy to any antibiotics
9. current alcohol or substance dependence

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Performance on Information Integration Learning Task | Testing Day (i.e. approx 3-5 hrs following placebo or D-cycloserine administration)
  Percent Correct Responses out of 240 trials (for schizophrenia patients) or 320 trials (for healthy adults) on the Information Integration Learning Task, which is a classification learning task in which participants learn to classify visual stimuli as category A or B following practice with stimuli and auditory feedback indicating correct versus incorrect responses.
Performance on Weather Prediction Learning Task | Testing Day (i.e. approx 3-5 hrs following placebo or D-cycloserine administration)
  Percent Correct Responses out of 240 trials (for schizophrenia patients) or 320 trials (for healthy adults) on the Weather Prediction Learning Task, which is a probabilistic classification learning task in which participants learn to predict the weather (i.e. "sun" or "rain" outcomes) based on combinations of cues that predict "sun" versus "rain" outcomes.
Performance on N-Back Working Memory Task | Testing Day (i.e. approx 3-5 hrs following placebo or D-cycloserine administration)
  Percent Correct Responses out of 240 trials (for schizophrenia patients) or 320 trials (for healthy adults) on the N-Back Task, which is a spatial working memory task in which participants identify whether each new stimulus on the computer screen is in the same location as the stimulus shown in trials ago. Patients with schizophrenia completed 80 trials at each of 3 working memory loads (0-, 1-, 2-back loads) and healthy adults completed 80 trials at each of 4 working memory loads (0-, 1-, 2-, 3-back loads).
Change in Visual Evoked Potential Amplitude using Electroencephalograph (EEG) | Testing Day (i.e. approx 3-5 hrs following placebo or D-cycloserine administration)
  EEG data were recorded using a 128 channel cap while participants viewed a black and white checkerboard stimulus on a computer screen in 6 x 2-minute blocks before and after viewing a quickly flashing checkerboard stimulus for 2 minutes. Change in the mean amplitude of the visual evoked potential from before versus after viewing the quickly flashing checkerboard stimulus was used to assess plasticity.

IPD SHARING:
Plan to Share IPD: Undecided